CLINICAL TRIAL: NCT02225015
Title: Cancer Prevention in Women With a BRCA Mutation: A Follow-up Genetic Counselling Intervention
Brief Title: Cancer Prevention in Women With a BRCA Mutation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women's College Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); London Health Sciences Centre (Other); Princess Margaret Hospital, Canada (Other); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 324638
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: BRCA1 Gene Mutation; BRCA2 Gene Mutation; Breast Cancer; Ovarian Cancer
Keywords: Cancer; Breast cancer; Ovarian cancer; BRCA Mutation; BRCA1 Gene Mutation; BRCA2 Gene Mutation; Telephone genetic counselling; Cancer prevention
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FTGC at 1 month (Active Comparator): Individuals randomized to the intervention group will receive a tailored cancer risk assessment via a follow-up telephone genetic counselling (FTGC) session within one month of study enrollment.
  Interventions: Behavioral: Follow-up Telephone Genetic Counselling
- Standard Care + FTGC in 12 months (No Intervention): Individuals randomized to the intervention group will receive a tailored cancer risk assessment at 12 months following study enrollment

INTERVENTIONS:
Behavioral: Follow-up Telephone Genetic Counselling — Individualized theoretical genetic counselling among women with BRCA mutations to assess the impact it has on the uptake of cancer prevention strategies.
  Arms: FTGC at 1 month

SUMMARY:
This study aims to develop a follow-up telephone-based genetic counselling (FTGC) intervention for women with a BRCA1 or BRCA2 mutation who have received genetic counseling in the past. Typically, when women undergo genetic testing, they receive standard genetic counselling prior to testing in order to fully understand the procedure and associated implications. If a woman's genetic test results are positive for a mutation, cancer prevention options are then discussed with a counsellor. However, in Canada, there is currently no formal follow-up counselling for women with a BRCA mutation to provide ongoing guidance and support about latest risk reduction strategies. Standard care relies on women making contact for any follow-up questions or concerns they may have. As a result, these women might not have the most current information regarding genetic risk assessment and prevention options. Therefore, individuals are being asked to participate in this study to aid research about the efficacy of FTGC in women with a BRCA mutation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed BRCA mutation
* Age 35 to 70 years
* No previous bilateral salpingo-oophorectomy
* No previous or current ovarian cancer
* At least 12 months since genetic testing or most recent contact by Narod follow-up study
* Can speak and understand English

Exclusion Criteria:

* Currently receiving treatment for another cancer diagnosis
* Pregnant
* Given birth in the last 6 months
* Booked surgical date for BSO

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of FTGC session | 3 years
  The primary aim is to determine the effects of a tailored risk communication intervention (FTGC) compared to a standard intervention

SECONDARY OUTCOMES:
Emotional and cognitive outcomes of intervention | 3 yrs
  Secondary aims are to compare the two study groups with regard to intent of cancer prevention strategies, decisional conflict, cancer-related distress, cancer risk and prevention knowledge, choice predisposition and health service utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Metcalfe, Dr., Principal Investigator — University of Toronto
Locations (3):
- Canada (3):
  - London Regional Cancer Centre, London, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Background] Kinney AY, Boonyasiriwat W, Walters ST, Pappas LM, Stroup AM, Schwartz MD, Edwards SL, Rogers A, Kohlmann WK, Boucher KM, Vernon SW, Simmons RG, Lowery JT, Flores K, Wiggins CL, Hill DA, Burt RW, Williams MS, Higginbotham JC. Telehealth personalized cancer risk communication to motivate colonoscopy in relatives of patients with colorectal cancer: the family CARE Randomized controlled trial. J Clin Oncol. 2014 Mar 1;32(7):654-62. doi: 10.1200/JCO.2013.51.6765. Epub 2014 Jan 21. PMID 24449229
- [Background] Kauff ND, Domchek SM, Friebel TM, Robson ME, Lee J, Garber JE, Isaacs C, Evans DG, Lynch H, Eeles RA, Neuhausen SL, Daly MB, Matloff E, Blum JL, Sabbatini P, Barakat RR, Hudis C, Norton L, Offit K, Rebbeck TR. Risk-reducing salpingo-oophorectomy for the prevention of BRCA1- and BRCA2-associated breast and gynecologic cancer: a multicenter, prospective study. J Clin Oncol. 2008 Mar 10;26(8):1331-7. doi: 10.1200/JCO.2007.13.9626. Epub 2008 Feb 11. PMID 18268356
- [Background] Rebbeck TR, Lynch HT, Neuhausen SL, Narod SA, Van't Veer L, Garber JE, Evans G, Isaacs C, Daly MB, Matloff E, Olopade OI, Weber BL; Prevention and Observation of Surgical End Points Study Group. Prophylactic oophorectomy in carriers of BRCA1 or BRCA2 mutations. N Engl J Med. 2002 May 23;346(21):1616-22. doi: 10.1056/NEJMoa012158. Epub 2002 May 20. PMID 12023993